CLINICAL TRIAL: NCT07318610
Title: A Master Protocol for a Phase 3, Multicenter, Randomized Study to Evaluate the Efficacy and Safety of REGN7508 and REGN9933, Monoclonal Antibodies Against Factor XI, in Participants With Recent Lower Extremity Revascularization for Symptomatic Peripheral Artery Disease (ROXI-PALISADE)
Brief Title: Reducing Adverse Vascular Outcomes With Factor XI Inhibition in Adult Participants With Peripheral Artery Disease
Acronym: ROXI-PALISADE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R9933-PAD-2394; 2025-522954-37-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Blood clots; Lower Extremity Revascularization (LER)
MeSH Terms: conditions — Peripheral Arterial Disease; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort 1 of this study is double-blinded, and for Cohort 2 the participants, sponsor, and the investigators will be blinded to REGN7508 or REGN9933, but rivaroxaban will be administered as open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: REGN7508; Drug: REGN9933; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: REGN7508; Drug: REGN9933; Drug: Rivaroxaban

INTERVENTIONS:
Drug: REGN7508 — Administered per the protocol
Drug: REGN9933 — Administered per the protocol
Drug: Placebo — Administered per the protocol
  Arms: Cohort 1
Drug: Rivaroxaban — Administered per the protocol
  Arms: Cohort 2

SUMMARY:
This study is researching 2 different experimental drugs called REGN7508 and REGN9933. The study is focused on people who have Peripheral Artery Disease (PAD), which means that the blood vessels in their arms and legs have become too narrow. People with PAD have a higher risk of getting blood clots after procedures like Lower Extremity Revascularization (LER), a procedure to improve blood flow in the legs and feet.

The aim of this study is to see how well REGN7508 and REGN9933 prevent life-threatening blood clots in participants with PAD who have recently had LER. The effects of REGN7508 and REGN9933, individually, will also be compared to rivaroxaban and a placebo.

The study is looking at several other research questions, including:

* What side effects might happen from taking the study drugs and how do they compare to the side effects of rivaroxaban
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drugs (which could make the drugs less effective or could lead to side effects)
* If the study drugs affect the ability of the blood to clot normally

ELIGIBILITY:
Key Inclusion Criteria:

1. Successful LER distal to the external iliac artery for ischemia due to atherosclerotic disease within 10 days prior to randomization as described in the protocol
2. At least 1 enrichment factor for major thrombotic vascular events:

   1. Bypass with prosthetic graft
   2. Endovascular treatment with stenting
   3. Target lesion length >15 cm
   4. History of LER or amputation for PAD prior to qualifying LER
   5. Type 2 diabetes mellitus requiring treatment
   6. Comorbid symptomatic coronary artery disease as described in the protocol
   7. Chronic kidney disease as described in the protocol
   8. Age ≥75 years

Key Exclusion Criteria:

1. Has any active clinical condition requiring therapeutic anticoagulation after the index revascularization including known triple positive antiphospholipid syndrome
2. Has known bleeding diathesis, platelet count <50,000/mm^3 or history of non-traumatic intracerebral hemorrhage, known cerebral amyloid angiopathy, or known unrepaired cerebrovascular malformations
3. Has recent coronary revascularization as described in the protocol
4. For Cohort 2 only: Has Glomerular Filtration Rate (GFR) <15 mL/min/1.73m^2 within 14 days prior to randomization or on dialysis or expected to be started on dialysis within the next 12 weeks starting from randomization
5. Has any other condition or therapy which would make the participant unsuitable for this study or not allow participation for the full planned study period
6. Has allergy, hypersensitivity, or other contraindication to REGN7508, REGN9933, or rivaroxaban (Cohort 2 only) or their excipients

Note: Other Protocol Defined Inclusion/ Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7050 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-05-05 (Estimated); Study Completion 2029-08-03 (Estimated)

PRIMARY OUTCOMES:
Time-to-first occurrence of a major thrombotic vascular event, consisting of Acute Limb Ischemia (ALI), major amputation (above the ankle) of vascular etiology, Myocardial Infarction (MI), ischemic stroke, or Cardiovascular (CV) death | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of International Society of Thrombosis and Hemostasis (ISTH) major or Clinically Relevant Non-major (CRNM) bleeding | Approximately up to 42 months
  Cohort 1 and 2

SECONDARY OUTCOMES:
Total (first and subsequent) occurrences of major thrombotic vascular events, consisting of ALI, major amputation (above the ankle) of vascular etiology, MI, ischemic stroke, or CV death | Approximately up to 42 months
  Cohort 1 and 2
Time-to-first occurrence of an expanded thrombotic vascular event, consisting of ALI, major amputation (above the ankle) of vascular etiology, MI, ischemic stroke, CV death, unplanned index limb revascularization, or Venous Thromboembolism (VTE) | Approximately up to 42 months
  Cohort 1 and 2
Time-to-first occurrence of ALI, major amputation (above the ankle) of vascular etiology, MI, ischemic stroke or coronary death | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of vascular hospitalization for a coronary or peripheral event of thrombotic nature | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of ALI, major amputation of vascular etiology, MI, ischemic stroke, or all-cause mortality | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of unplanned index limb revascularization for ischemia | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of VTE | Approximately up to 42 months
  Cohort 1
Time-to-all-cause mortality | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of Major Adverse Limb Event (MALE) | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of Major Adverse Cardiovascular Event (MACE) | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of a major thrombotic vascular event or ISTH fatal/critical organ bleeding (net clinical benefit) | Approximately up to 42 months
  Cohort 1
Time-to-first occurrence of Thrombolysis in Myocardial Infarction (TIMI) major bleeding | Approximately up to 42 months
  Cohort 1 and 2
Occurrence of Treatment-Emergent Adverse Event (TEAEs) | Approximately up to 45 months
  Cohort 1 and 2
Severity of TEAEs | Approximately up to 45 months
  Cohort 1 and 2
Occurrence of Anti-Drug Antibody (ADA) to REGN7508 over time | Approximately up to 45 months
  Cohort 1 and 2
Magnitude of ADA to REGN7508 over time | Approximately up to 45 months
  Cohort 1 and 2
Occurrence of ADA to REGN9933 over time | Approximately up to 45 months
  Cohort 1 and 2
Magnitude of ADA to REGN9933 over time | Approximately up to 45 months
  Cohort 1 and 2
Concentrations of REGN7508 over time | Approximately up to 45 months
  Cohort 1 and 2
Concentrations of REGN9933 over time | Approximately up to 45 months
  Cohort 1 and 2
Change from baseline in activated Partial Thromboplastin Time (aPTT) over time | Approximately up to week 9
  Cohort 1 and 2
Change from baseline in Prothrombin Time (PT)/International Normalization Ratio (INR) over time | Approximately up to week 9
  Cohort 1 and 2
Total (first and subsequent) occurrences of expanded thrombotic vascular events | Approximately up to 42 months
  Cohort 2
Time-to-first occurrence of a major thrombotic vascular event | Approximately up to 42 months
  Cohort 2
Total (first and subsequent) occurrences of ALI, major amputation (above the ankle) of vascular etiology, MI, all-cause stroke, or CV death | Approximately up to 42 months
  Cohort 2
Total (first and subsequent) occurrences of ALI, major amputation (above the ankle) of vascular etiology, MI, all-cause stroke, CV death, unplanned index limb revascularization, or VTE | Approximately up to 42 months
  Cohort 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/